CLINICAL TRIAL: NCT01019226
Title: Implementation of Work in Progress (WIP) Sequences in MRI
Brief Title: Implementation of Work in Progress (WIP) Sequences in Magnetic Resonance Imaging (MRI)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sheba Medical Center, Sheba Medical Center
Other Study IDs: SHEBA-09-7000-EK-CTIL
Record Dates: First submitted 2009-11-22; First posted 2009-11-25 (Estimated); Last update posted 2010-05-11 (Estimated); Status verified 2010-05

CONDITIONS: Ischemic Cardiomyopathy; Nonischemic Cardiomyopathy
Keywords: myocardium; Magnetic resonance imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- cardiac MRI: Ischemic cardiomyopathy, non ischemic cardiomyopathy, myocarditis, cardiomyopathy

SUMMARY:
Trial of new work in progress (WIP) sequences in MRI.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of ischemic or non ischemic cardiomyopathy

Exclusion Criteria:

* claustrophobia
* irregular heart rhythm

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cardiac MRI
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2009-12; Primary Completion 2011-05 (Estimated); Study Completion 2011-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Eli Konen, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba medical center, Tel Litwinsky, Israel